CLINICAL TRIAL: NCT00311064
Title: Inflammatory Response and Pregnancy Outcome in Women With Type 2 Diabetes or Only Overweight. The Influence of Physical Activity
Brief Title: Inflammatory Response and Pregnancy Outcome in Women With Type 2 Diabetes or Overweight
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: because of lack of funding and recruitment problems the study has been closed.
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 01 285157
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Exercise

INTERVENTIONS:
Behavioral: physical activity

SUMMARY:
Purpose:

The purpose of this study is to determine if disturbances in cytokines or factors of the metabolic syndrome, can predict complications in pregnancy, birth, and the perinatal period in pregnant women with type 2 diabetes or who are overweight. At the same time we, the investigators at Rigshospitalet, want to determine if physical activity in the overweight pregnant woman can influence these factors in a favourable way and, with that, improve the progress of pregnancy and birth.

DETAILED DESCRIPTION:
Material and Method:

This study falls in two fields:

First 80 pregnant women with type 2 diabetes are followed with determination of cytokines and factors of the metabolic syndrome throughout the pregnancy. The correlation between these variables and the pregnancy and delivery progress is evaluated.

280 overweight (body mass index [BMI] > 30 kg/m2) pregnant women with no medical conditions are examined in the same way. The women are randomized in week 14 to either continue their habitual physical activity or to elevate it by participating in a training program with other pregnant women 3 times weekly.

Both groups will get blood samples taken during fasting approximately 50 ml 3-4 times during the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* BMI < 45 kg/m2
* Healthy
* Over 18 years of age
* No earlier preterm delivery (before 37)
* Singleton pregnancy
* 14 weeks +/- 1 week of gestation

Exclusion Criteria:

* BMI > 45 kg/m2
* Earlier preterm delivery (before 37)
* Not singleton pregnancy
* Medically treated diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2006-03; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
perinatal mortality
congenital malformations and preeclampsia
gestational hypertension and gestational diabetes mellitus (GDM)
preterm delivery
too large infants (> 2 standard deviation [SD])

SECONDARY OUTCOMES:
delivery by caesarian section
induction of labour

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Breitowicz, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Obstetric Clinic, Juliane Marie Centret, Copenhagen, Østerbro, Denmark